CLINICAL TRIAL: NCT00997282
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, 3-arms Parallel Group Comparative Study of OPC-262 in Patients With Type 2 Diabetes (Phase 2/3 Study)
Brief Title: A Study of OPC-262 in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Katsuhisa Saito, Senior Operating Officer, Department of Clinical Research and Development, Otsuka Pharmaceutical Co., Ltd.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 262-09-001; JapicCTI-090904
Record Dates: First submitted 2009-10-16; First posted 2009-10-19 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Diabetes Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- OPC-262 2.5 mg (Experimental): orally administered once daily for 24 weeks
  Interventions: Drug: OPC-262 2.5 mg
- OPC-262 5 mg (Experimental): orally administered once daily for 24 weeks
  Interventions: Drug: OPC-262 5 mg
- Placebo (Placebo Comparator): orally administered once daily for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OPC-262 2.5 mg — orally administered once daily for 24 weeks
  Arms: OPC-262 2.5 mg
Drug: OPC-262 5 mg — orally administered once daily for 24 weeks
  Arms: OPC-262 5 mg
Drug: Placebo — orally administered once daily for 24 weeks
  Arms: Placebo

SUMMARY:
The purpose of this clinical study is to evaluate the superiority of the efficacy of OPC-262 (2.5 mg, and 5 mg) to placebo in patients with type 2 diabetes after 24 week treatment in a double-blind fashion and to evaluate the safety of OPC-262 to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes patients with HbA1C above 6.5% and below 10%
2. Patients who are capable of giving informed consent
3. Patients who are able to take contraceptive measures to avoid pregnancy of the patient or the patient's partner for the entire study period and for 4 weeks after the study (end of the post-observation period)

Exclusion Criteria:

1. Patients with type 1 diabetes mellitus, patients with diabetes mellitus due to other specified drugs, mechanisms or diseases, and patients with gestational diabetes mellitus
2. Patients with a medical history of diabetic coma
3. Patients with poorly-controlled hypertension
4. Patients with heart failure
5. Patients with a complication of active hepatitis or hepatic cirrhosis
6. Patients undergoing treatment of glomerular diseases other than diabetic nephropathy
7. Patients with a history or complication of malignant tumor

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Changes in HbA1C from baseline | Week 24 (LOCF)

SECONDARY OUTCOMES:
Changes in fasting blood glucose (FBG) from baseline | Week 24
Changes in 2 hour postprandial blood glucose (PPG) from baseline | Week 24
Changes in 3 hour PPG AUC from baseline | Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Kaatsuhisa Saito, Study Chair — OPCJ
Locations (7):
- Japan (7):
  - Chubu Region
  - Chugoku Region
  - Kansai Region
  - Kanto Region
  - Kyushu Region
  - Shikoku Region
  - Tohoku Region